CLINICAL TRIAL: NCT06349629
Title: The Clinical Study of 3D-printed Magnesium Alloy Prosthesis With Controllable Degradation Rate in the Repair of Periarticular Bone Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Tian Yun, Professor, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240401
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Degradation of Magnesium Alloy Prosthesis and New Bone Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical effect of 3D printed magnesium alloy prosthesis for repairing proximal humerus bone defect. (Experimental): The 3D printed magnesium alloy prosthesis is used to repair the proximal humerus fracture with bone defect, and the dynamic process of prosthesis degradation, fracture healing and new bone growth will be observed.
  Interventions: Device: 3D printed WE43 magnesium alloy
- Clinical effect of 3D printed magnesium alloy prosthesis for repairing distal radius bone defect. (Experimental): The 3D printed magnesium alloy prosthesis is used to repair the distal radius fracture with bone defect, and the dynamic process of prosthesis degradation, fracture healing and new bone growth will be observed.
  Interventions: Device: 3D printed WE43 magnesium alloy
- Clinical effect of 3D printed magnesium alloy prosthesis for repairing tibial plateau bone defect. (Experimental): The 3D printed magnesium alloy prosthesis is used to repair the tibial plateau fracture with bone defect, and the dynamic process of prosthesis degradation, fracture healing and new bone growth will be observed.
  Interventions: Device: 3D printed WE43 magnesium alloy

INTERVENTIONS:
Device: 3D printed WE43 magnesium alloy — This 3D printed WE43 magnesium alloy has porous structure and suitable mechanical strength, can be stable in the bone support, and gradually degrade to promote bone healing.

SUMMARY:
Perimarticular fracture bone defect is a common and complicated clinical disease. The current treatment for this type of injury is anatomical reduction of the fracture, where the bone defect is filled with artificial, autologous or allogeneic bone in granular form, and then fixed with plates and screws. However, these bone filler materials exist in a loose accumulation state and cannot form an effective overall support force for the joint. The applicant realized three dimensional (3D) printing of WE43 magnesium alloy with personalized design and porous overall structure, and developed high-temperature heat treatment technology to slow its degradation, which effectively realized the dual stability of degradation rate of magnesium alloy support body and overall structure during the bone repair period. This project will optimize the design of 3D printed WE43 magnesium alloy full-structure in-bone support, and establish a metamaterial pore structure design platform that regulates the physical properties and degradation behavior of porous implants. Fracture from proximal humerus, distal radius and tibial plateau

ELIGIBILITY:
Inclusion Criteria:

1. Patients with traumatic periarticular fractures of extremities with bone defects requiring bone grafting mainly include distal radius fractures, proximal humerus fractures, and tibial plateau fractures.
2. Between the ages of 18 and 70.
3. Sign informed consent, voluntarily participate in the study, and complete postoperative follow-up.
4. There are no obvious surgical contraindications and no contraindications for magnesium alloy prosthesis implantation.

Exclusion Criteria:

* Patients with pathological fracture ② pregnant women ③ doctors evaluated other conditions that were not suitable for inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Magnesium alloy metabolism | 1, 3, 6, 12, 24 months after surgery
  Blood routine, electrolyte, liver and kidney function, urine routine were used to evaluate magnesium alloy metabolism in vivo.
Degradation of 3D printed magnesium alloy prosthesis | 1, 3, 6, 12, 24 months after surgery
  X-ray and computed tomography (CT) scans were used to evaluate the degradation progression of 3D printed magnesium alloy prosthesis
New bone regeneration | 1, 3, 6, 12, 24 months after surgery
  X-ray and CT scans were used to evaluate the process of new bone regeneration
Evaluation of shoulder joint function | 1, 3, 6, 12, 24 months after surgery
  American Shoulder and Elbow Surgeon's Form (ASES) was used to evaluate the shoulder joint function. The score scale of this form was 0 to 100, higher score represents better shoulder joint function.
Evaluation of wrist joint function | 1, 3, 6, 12, 24 months after surgery
  Mayo Wrist Score was used to evaluate the wrist joint function.The score scale of this form was 0 to 100, higher score represents better joint function.
Evaluation of knee joint function | 1, 3, 6, 12, 24 months after surgery
  Knee Society Score (KSS) was used to evaluate the knee joint function.The score scale of this form was 0 to 100, higher score represents better joint function.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Haidian
  - Peking University Third Hospita, Beijing